CLINICAL TRIAL: NCT00008697
Title: A Phase I/II Trial of Infusional Arsenic Trioxide for Relapsed Acute Promyelocytic Leukemia
Brief Title: Arsenic Trioxide in Treating Patients With Refractory or Recurrent Acute Promyelocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: CDR0000066617; WU-98-0185; NCI-V98-1466
Record Dates: First submitted 2001-01-13; First posted 2003-01-27 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Leukemia
Keywords: recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; adult acute promyelocytic leukemia (M3); childhood acute promyelocytic leukemia (M3)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1 (Experimental): Cohort 1 Arsenic trioxide = 0.1 mg/kg/day x 28 days with 14 day rest for 3 cycles (each cycle = 6 weeks)
  Cohort 2 Arsenic trioxide = 0.15 mg/kg/day x 28 days with 14 day rest for 3 cycles (each cycle = 6 weeks)
  Cohort 3 Arsenic trioxide = 0.20 mg/kg/day x 28 days with 14 day rest for 3 cycles (each cycle = 6 weeks)
  Cohort 4 Arsenic trioxide = 0.25 mg/kg/day x 28 days with 14 day rest for 3 cycles (each cycle = 6 weeks)
  Cohort 5 Arsenic trioxide = 0.30 mg/kg/day x 28 days with 14 day rest for 3 cycles (each cycle = 6 weeks)
  Interventions: Drug: arsenic trioxide
- Phase 2 (Experimental): Arsenic trioxide = MTD found in Phase 1 mg/kg/day x 28 days with 14 day rest for 3 cycles (each cycle = 6 weeks)
  Interventions: Drug: arsenic trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
The purpose of this study is to evaluate both the efficacy and toxicity of infusional arsenic trioxide in the treatment of patients with relapsed or refractory acute promyelocytic leukemia (APML). In addition, correlation between pharmacokinetic data and both therapeutic response and therapy-related toxicities will be sought.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study.

Patients receive arsenic trioxide IV over 2 hours daily for 28 days followed by a 14 day rest period. Patients may receive up to 3 courses of treatment.

Dose escalation continues in cohorts of 3-6 patients until the maximum tolerated dose (MTD) or minimum effective dose (MED) is determined. The MTD is defined as the dose preceding that at which 2 or more patients experience dose limiting toxicity. The MED is defined as the dose at which 4 of 6 patients achieve a complete cytogenetic or molecular response. After the MTD or MED is determined, an additional 20 patients are enrolled at this dose level.

Patients are followed monthly for 6 months and every three months for an additional 1.5 years.

ELIGIBILITY:
INCLUSION CRITERIA

1. APML diagnosis based upon morphological, histochemical, and/or flow cytometric criteria, confirmed upon review by a central, study-designated hematologic pathologist;

   OR

   any relapsed acute leukemia bearing a t(15:17) translocation or variant APML translocations involving the retinoic acid receptor alpha gene on chromosome 15q22, based on cytogenetics or PCR.
2. disease in first or subsequent relapse, following standard induction and consolidation chemotherapy (with all-trans retinoic acid) and/or allogeneic bone marrow/stem cell transplantation;

OR

failure to achieve initial complete remission with ATRA and standard chemotherapy.

EXCLUSION CRITERIA

1. Availability of a fully HLA-matched sibling donor for patients otherwise felt to be candidates for allogeneic bone marrow/stem cell transplantation; patients with only a partially HLA-matched sibling or matched unrelated donor will remain eligible for study entry.
2. pregnancy.
3. Patients with significantly impaired left ventricular ejection fraction (<40%) will be ineligible for the study.

Patients with renal failure and a creatinine clearance of less than 25 ml/min or requiring hemodialysis will be ineligible for the study. Otherwise, there are no rigid exclusion criteria based upon age, performance status, or co-morbidity. Decisions regarding enrollment of patients for whom these factors may be relevant will be individualized and left to the discretion of the investigators. Central venous access will be required for all patients. Patients of child-bearing potential must agree to use contraception during sexual intercourse while undergoing treatment with arsenic trioxide.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1998-11; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) or minimum effective dose (MED) | 6 weeks
Efficacy (response and survival) at the MTD - Phase 2 only | 18 weeks

SECONDARY OUTCOMES:
Acute and chronic toxicities | 18 weeks
Evaluation of the pharmacokinetics and their correlation with toxicities and response | 18 weeks
Evaluation of PML/RARA and PML protein redistribution and degradation following treatment and their correlation with response | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John F. DiPersio, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States